CLINICAL TRIAL: NCT02616575
Title: The Application of Smart Health Management System on Home-Care for Elderly Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201502062RINB
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Peer Review, Health Care
Keywords: home care; monitoring system; risk assessment; telehealth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Silver link: Patients enrolled in NTUH hospital and its Behui branch

SUMMARY:
Aims: The purposes of this study are

1. to create a smart living environment with home care system using GPS and cloud-based services for elderly people.
2. to improve the home care system from user feedback and recommendations.

Methods: Participants (n = 50) will be recruited from geriatric clinics in National Taiwan University Hospital (NTUH) main hospital and its Beihu branch. Enrollment criteria include: aged 60 or older, living alone or with one companion (not children), taking at least one chronic medications, having the capability to understand the study and complete the study, willing to participate into the study with telephone follow ups.

DETAILED DESCRIPTION:
Background: At present, with the changing of the society structure, the ratio of nuclear family and older people who live alone is arising. Therefore, making care system fit for aging population to create a appropriate healthcare is cricial. Thus, the investigators have established a smart home health care system, SilverLink to improve resident quality for older adults living alone.

Aims: The purposes of this study are

1. to create a smart living environment with home care system using GPS and cloud-based services for elderly people.
2. to improve the home care system from user feedback and recommendations.

Methods: Participants (n = 50) will be recruited from geriatric clinics in NTUH main hospital and its Beihu branch. Enrollment criteria include: aged 60 or older, living alone or with a companion (not children), taking at least one chronic medications, having the capability to understand the study and complete the study, willing to participate into the study with telephone follow ups.

This study includes two sessions:

1. set up the healthcare system, with home GPS and sensors. The investigators will stick small sensors on fridge door, pillbox, pendant…for automatic detection of the frequency of food intake, take medicine and get out of home….Also, the investigators will use accelerometer to track the body movement for older adults.
2. use APP for blood pressure (BP) or other measurements data tracking. The investigators develop an APP system to help older adults to log in and track their dairy physiological measurements. (optional)

Anticipated results:

Provide feasibility data for system to allow future modifications of the system.

Improve older adults' life quality and satisfaction. Under the integration of this healthcare technology and the central communication medical services may create a smart healthcare network, which is not only the effectiveness on reducing medical costs, but also will provide a convenient connection between living alone older adults and their family.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 or older,
* living alone or with a companion (not children),
* taking at least one chronic medications,
* having the capability to understand the study and complete the study,
* willing to participate into the study with telephone follow ups.

Exclusion Criteria:

* If patients were unable to meet at least the inclusion criteria above.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: aged 60 or older, living alone or with a companion (not children), taking at least one chronic medications, having the capability to understand the study and complete the study, willing to participate into the study with telephone follow ups.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-12; Primary Completion 2021-03 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | 3 months
  We developed a self-completed, 23-item questionnaire, 5-point Likert scale, ranging from 1 (very satisfied) to 5 (very dissatisfied) for the purpose of how patient feel about this Silverlink system and the online website.,

SECONDARY OUTCOMES:
Medication adherence | 3 months
  defined as number of pill box opened/ expected number of pill box to be opened in past 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ding-Cheng Chan, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan